CLINICAL TRIAL: NCT02426957
Title: Brief Alcohol Intervention for Adolescents Who Have Attempted Suicide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Kimberly H. McManama O'Brien, Researcher, Boston Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: A00013929
Record Dates: First submitted 2015-03-26; First posted 2015-04-27 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Suicide; Alcohol Drinking
MeSH Terms: conditions — Suicide; Alcohol Drinking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Enhancement Therapy (Experimental): The 60-90 minute intervention consists of the following components: establishing rapport, assessing motivation for change, enhancing motivation for change, envisioning the future, establishing goals, and completing goals, strategies, and change plan worksheets. Personalized feedback for the intervention will be derived from the assessment battery and will be provided in both written and graphic formats. In addition to the 60-90 minute MI intervention delivered to the adolescent, a 30-45 minute intervention will be conducted with the adolescent and parent(s) the following day, in which the adolescent will review the goals, strategies, and change plan worksheets with the parent(s), facilitated by the therapist.
  Interventions: Behavioral: motivational enhancement therapy
- Treatment As Usual (No Intervention): Treatment As Usual on inpatient psychiatric unit

INTERVENTIONS:
Behavioral: motivational enhancement therapy — The intervention consists of the following components: establishing rapport, assessing motivation for change, enhancing motivation for change, envisioning the future, establishing goals, and completing goals, strategies, and change plan worksheets.
  Arms: Motivational Enhancement Therapy

SUMMARY:
The study will use a two group randomized controlled trial to compare a brief motivational interviewing (MI) intervention to TAU with 50 adolescents psychiatrically hospitalized for a suicide plan or attempt who have co-occurring alcohol use. Data will be collected via in-person interviews and self-administered questionnaires at baseline and 3 month follow-up assessments to explore outcome changes in negative alcohol expectancies, confidence in ability to handle situations where alcohol is present, likelihood of receiving alcohol treatment, frequency of alcohol use, and suicidal ideation, suicide planning, and suicide attempts for adolescents receiving the intervention relative to TAU.

DETAILED DESCRIPTION:
A two group randomized controlled trial will be used to compare the brief MI intervention to TAU with 50 adolescents psychiatrically hospitalized for a suicide plan or attempt who have co-occurring alcohol use. Adolescents admitted to the unit for a suicide plan or attempt will be screened by PI O'Brien or Co-I White within 24 hours of their admission to determine if they meet criteria for alcohol use in past month by selecting 1-6 on Question #1 of the Adolescent Drinking Questionnaire (ADQ). Then Co-I White (or PI O'Brien in the event Co-I White is unavailable) will administer the Drug Use Questionnaire (DUQ), Timeline Follow-back Interview (TLFB), Brief Situational Confidence Questionnaire (BSCQ), Comprehensive Effects of Alcohol (CEOA), Opinions About Alcohol Use (OAAU), Suicide Ideation Questionnaire (SIQ), Inventory of Motivations for Suicide Attempts (IMSA), and a subset of questions from the Columbia-Suicide Severity Rating Scale (C-SSRS). Once assessment measures are completed, participants will be randomized to either the experimental condition or TAU. Randomization will be accomplished by using an urn randomization procedure used to retain random allocation while balancing relative probabilities of assignment to treatment groups. Urn randomization in contrast to simple or block randomization is dynamic; the probability of treatment assignment changes dependent on the degree of treatment imbalance throughout the course of the trial. We will randomize by 1) ADQ score (i.e., adolescents scoring <4 which indicates drinking at least 2-3 times per week) and 2) gender. The adolescent will receive the individual MI intervention in a private room on the inpatient psychiatric unit; the family intervention will be delivered in a private room on the unit, ideally the next day. After the intervention the adolescent will complete the exit interview and Session Evaluation Form (SEF) to assess acceptability. Once a discharge date is made for the participant, PI O'Brien or Co-I White will schedule a 3 month follow-up appointments with the adolescent and guardian; the ADQ, DUQ, TLFB, BSCQ, CEOA, SIQ, IMSA, and C-SSRS will be readministered at the follow-up assessment in a private room in the visitors' area of the inpatient psychiatric unit by RA Wigglesworth, so that the clinician conducting the assessment is blind to condition.

ELIGIBILITY:
Inclusion Criteria:

* current hospitalization for suicide plan or attempt,
* alcohol use in past month, indicated by selecting 1-6 on Question #1 of the Adolescent Drinking Questionnaire (ADQ) which is currently given to all patients to fill out upon admission to the inpatient psychiatric unit,
* age 13-17, and 4) ability to communicate in English.

Exclusion Criteria:

* developmental delay, autism spectrum disorder, or psychosis, per chart review.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
alcohol use | 3 months
  Adolescent Drinking Questionnaire (ADQ). The ADQ is a 6 item self-report measure assessing drinking frequency (days per month), quantity (drinks per occasion), frequency of high-volume drinking (≥ 5 drinks per occasion), and frequency of intoxication (feeling "drunk" or "very, very high"), over the past month.
  Timeline Follow-back Interview (TLFB). The TLFB is a widely-used research and clinical assessment tool with good reliability and validity for various groups of individuals with alcohol use problems. The TLFB collects alcohol and drug consumption information using a calendar format with temporal cues to assist in recall of days when alcohol and drugs were used, and can be used to simultaneously recall other behaviors, such as suicidal ideation and attempts. The TLFB will be conducted using the prior 30 days at baseline and each follow-up.

SECONDARY OUTCOMES:
suicidal ideation | 3 months
  Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS assesses the range of suicidal behavior including preparatory acts, aborted attempt and interrupted attempt, and passive and active suicidal ideation, as well as intensity of ideation. To avoid redundancies in measures, we will not administer the intensity of ideation section to the participant, as some of that construct is captured by the SIQ. At follow-up, suicidality will be assessed only since the last assessment.
  Suicide Ideation Questionnaire (SIQ). The SIQ is a 30 item self-report instrument that assesses suicidal ideation in adolescents over the past month. Items are rated on a 7-point Likert scale (0=I never had this thought, to 6=almost every day). Coefficient alpha internal consistency measures for the SIQ have been reported at 0.97 as well as good construct validity.

OTHER OUTCOMES:
drug use | 3 months
  Drug Use Questionnaire (DUQ). The DUQ assesses the number of days adolescents used substances over the past 30 days including nicotine, marijuana, cocaine, LSD, PCP, inhalants, etc. Internal consistency in one study sample was .75 (alpha = .80 when inhalants was dropped). Test/retest for mean number of days each substance was used was .83 from 3 to 6 month follow-up and .94 from 6 to 12 month follow-up.
situational confidence | 3 months
  Brief Situational Confidence Questionnaire (BSCQ). The BSCQ is an eight item self-report instrument used to assess confidence in one's ability to resist the urge to use alcohol or other substances. Responses are provided on 10-point Likert scales (i.e., 10% increments, from 0%=not at all confident to 100%=completely confident). The Cronbach's alpha coefficient was 0.85 in one study.
effects of alcohol | 3 months
  Comprehensive Effects of Alcohol (CEOA). The CEOA is 38 items and assesses positive and negative expected effects of alcohol and has demonstrated adequate internal consistency, temporal stability and construct validity.
opinions about alcohol | 3 months
  Opinions About Alcohol Use (OAAU). The OAAU is a two item self-report measure assessing the importance and confidence in reducing alcohol use. In addition to baseline and 3 month follow-up, this measure will be administered post-intervention to all participants randomized to the intervention, to assess for within session changes.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O'Brien, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided